CLINICAL TRIAL: NCT03215355
Title: Improving Cone-beam Computed Tomography for Image Guided Stereotactic Body Radiation Therapy of the Liver Using Gadoxetate Disodium
Brief Title: Improving CBCT for Liver IG-SBRT Using Gadoxetate Disodium
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Not approved
Sponsor: Slawa Cwajna (Other)
Collaborators: Nova Scotia Health Authority (Other)
Responsible Party: Sponsor-Investigator, Slawa Cwajna, Radiation Oncologist (MD), Nova Scotia Health Authority
Organization: Nova Scotia Health Authority (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NSHAREB#4793
Record Dates: First submitted 2017-07-05; First posted 2017-07-12 (Actual); Last update posted 2021-01-27 (Actual); Status verified 2021-01

CONDITIONS: Primary Liver Cancer; Metastatic Liver Cancer
Keywords: Adaptive radiotherapy; Contrast media; Cone-beam computed tomography; Stereotactic body radiation therapy
MeSH Terms: conditions — Carcinoma, Hepatocellular; Liver Neoplasms | interventions — gadolinium ethoxybenzyl DTPA

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Participants receiving Primovist (Experimental): Because this is a proof of concept study, only one arm will be considered which is the patients that receive the one time contrast injection prior to their first treatment. The intervention is that although this drug is approved, an off label dosing regiment is being used to improve a separate imaging modality than what it was approved for. Based on preliminary phantom experiments and toxicity results in the literature, four times the dose was deemed safe and required to use for CBCT.
  Interventions: Drug: Primovist

INTERVENTIONS:
Drug: Primovist — Primovist is currently a drug marketed for MRI. In this study it will be administered intravenously at 4 times what it is quoted for MRI to enhance the different imaging modality (CBCT) to improve the accuracy of liver SBRT. Although liver SBRT usually consists of 5 treatments, contrast will only be administered during the first treatment.
  Consulting Health Canada and Bayer HealthCare Canada (the drug manufacturer) deemed this use "off label dosing" which in Canada is at the discretion of the physician. Based on preliminary imaging testing, and a review of toxicity literature for this drug, the administration for this specific use was deemed appropriate to give adequate image quality, while simultaneously maintaining patient safety.
  Other Names: Gadoxetate disodium; Gd-EoB-DTPA

SUMMARY:
This is a feasibility study requiring only three patients to serve as a proof of concept that gadoxetate disodium (a liver specific contrast agent) can be used to improve images taken just before liver SBRT treatments.

The hypothesis of this research is that if gadoxetate disodium improves image quality at the time of treatment, then it can be used for image guided radiotherapy (IGRT). Image guidance is the procedure where the 3D CT image that is used to plan a radiotherapy treatment, is aligned to a 3D image taken just before treatment. The better the alignment, the more accurate the treatment, which is crucial for high dose treatments such as SBRT.

This research is important for two main reasons. First, it is much less invasive than the standard of care which involves surgically implanting markers in the liver that can move over time. The benefit to harm ratio for surgery, compared to an injection, is much more dramatic. Furthermore, not all patients are surgical candidates, and therefore in those cases radiation oncologists must prescribed a larger area to treat to ensure that none of the cancerous region is missed. The drawback to this method is the irradiation of more normal tissue than necessary, which although deemed to have a greater benefit than harm, is not ideal. Secondly, this research has strong implications in the field of radiation oncology to move towards patient oriented radiotherapy treatments. If successful, radiation treatment to the liver could be performed in less treatments because of the confidence given to radiation oncologists of the cancer location; knowing exactly the healthy liver regions to avoid.

DETAILED DESCRIPTION:
Preliminary testing has already been performed and proves the notion that to achieve adequate image quality in a CT imaging phantom, at least 4 times the MRI administration dose would be required. These conclusions were supported qualitatively by a radiologist, radiation oncologist, and medical physicist, while also being backed up by quantitative measurement that has been accepted in the medical imaging literature. It is important for this work to first ensure that the imaging system is optimized, to have confidence that it will be successful for patients. Therefore before this study begins, substantial time and effort will be spent using phantoms and optimizing the imaging parameters and protocol.

The current procedure for a patient that presents with liver cancer begins with a referral from the patient's primary care physician for stereotactic body radiation therapy (SBRT). A radiation oncologist makes the decision whether the patient is suitable for SBRT.

If the patient is deemed acceptable by the radiation oncologist, the next step is to undergo diagnostic imaging so that the radiation oncologist can identify where exactly the disease is located, and start the SBRT plan. Using the diagnostic images, the radiation oncologist outlines the areas to treat, as well as the areas that they want to spare. This information is given to a physicist who then plans the optimal way of delivering radiation based on the oncologist's specifications. Once the plan is approved by the radiation oncologist, the patient can be treated.

At the time of treatment, the patient is placed in an immobilization device on a treatment couch by a radiation therapist. Once the patient is immobilized, an x-ray imaging system that is attached to the treatment machine extends out towards the patient. The machine performs a 180-degree rotation with continuous x-ray imaging. Once sufficient imaging has been performed, the therapists then align these images with the previous diagnostic CT image that was used to plan the radiation treatment. This alignment process tells the radiation therapists how much to adjust the patient on the treatment couch to ensure the most accurate treatment delivery. Once the patient is in the proper position, the radiation treatment is delivered and then the patient can leave.

The treatment procedure is then performed on five separate days each separated by 48 hours.

The proposed research follows the same procedure with addition of a contrast injection at the treatment stage. A consent form will be given to the patient entailing the purpose of this study. It will highlight the risks and benefits of receiving contrast prior to the radiation treatment, as well as a complete outline of the research. If the patient consents to receiving an intravenous contrast injection of gadoxetate disodium then the treatment procedure will change as follows:

Before the patient is placed in the immobilization device, a MRI technologist with experience giving gadoxetate disodium injections will give the prescribed injection according to the patient's body weight. After the injection is given, a liver SBRT trained radiation therapist will lead the patient to the treatment machine and set them up in the immobilization device as per standard treatments. The same time-of-treatment imaging will be performed, with the hypothesis that the image quality will improve because of the addition of the contrast agent. The contrast agent will only be administered at the first treatment because of the limited data on repeat injections of the drug in humans. Furthermore, for the first treatment when contrast is administered, a radiation oncologist, radiologist, medical physicist, MRI technologist, and three radiation therapists will attend.

The patient will then be monitored for another 30 minutes with support equipment ready in the rare event that a side effect occurs.

As per standard treatments, the radiation oncologist will follow up with patients at regular intervals during and after treatment, making sure to check with the patient for possible side effects of using the contrast agent.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years and over
* Not suitable for surgery or radio-frequency ablation (RFA).
* Histologic confirmation of cancer diagnosis and/or histologic confirmation of liver malignancy
* Meets criteria for oligometastasis (not more than 5 metastases in total, none larger than 5cm in diameter, no more than 3 in any one organ).
* Child-Pugh: A
* > 700cc uninvolved liver
* No limitation on the actual size of the tumor providing organ at risk (OAR) dose constraints can be met
* ECOG performance status 0-2
* Acceptable kidney and liver function : (AST/ALT/GGT, alkaline phosphate, total bilirubin, albumin), normal serum creatinine or Creatinine clearance > 60mL/min
* Life expectancy > 6 months
* No chemotherapy within 4 weeks
* Recurrence at the site of prior liver resection

Exclusion Criteria:

* Age less than 18 years
* Previous diagnosis of chronic sever renal insufficiency
* Previous diagnosis of acute renal failure
* Previous diagnosis of acute kidney injury
* Patients with biliary obstruction
* Impaired liver enzymes (>6x ULN)
* Platelets < 50 000
* < 700cc of normal liver
* Ongoing or planned chemotherapy
* Progressing extra-hepatic disease
* History of active hepatitis
* Significant comorbidities within previous 6 months (unstable angina, MI, ascites, coagulopathy)
* Prior radiotherapy to site/sites of progressive disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-08 (Estimated); Primary Completion 2018-08 (Estimated); Study Completion 2018-08 (Estimated)

PRIMARY OUTCOMES:
Improved image quality after injection as determined by contrast-to-background calculation and expert observation. | 12 months
  Images will be read by a radiologist and radiation oncologist to qualitatively assess whether or not image enhancement occurred. This will be compared to the quantitative standard of calculating the amount of contrast in the region that is to be enhanced, compared to the surrounding normal tissue (background). Adequate enhancement will be taken as contrast-to-background ratio greater than 1.

SECONDARY OUTCOMES:
Toxicity with "off label" dosing | 12 months
  Categorized as adverse reaction or no adverse reaction post monitoring.

CONTACTS AND LOCATIONS:
Overall Officials: Slawa Cwajna, MD, Principal Investigator — Nova Scotia Health Authority
Locations (1):
- Nova Scotia Cancer Centre, Halifax, Nova Scotia, Canada